CLINICAL TRIAL: NCT06137638
Title: A Placebo-controlled, Double-blind, Randomized Trial to Evaluate the Efficacy of ENA-001 in Preventing Postoperative Respiratory Depression
Brief Title: ENA-001 for Post Operative Respiratory Depression (PORD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enalare Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ENA-001-201
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENA-001 Treatment Arm (Experimental): ENA-001 consisting of continuous infusion of a loading dose of 2.0 mg/kg/hr for 20 minutes followed by a maintenance dose of 1.1 mg/kg/hr.
  Interventions: Drug: ENA-001
- Placebo Treatment Arm (Placebo Comparator): Matching placebo for ENA-001 will consist of the solution that is used as diluent for ENA-001. Placebo will be administered similarly consisting of continuous infusion of a loading dose of 2.0 mg/kg/hr for 20 minutes followed by a maintenance dose of 1.1 mg/kg/hr.
  Interventions: Drug: ENA-001

INTERVENTIONS:
Drug: ENA-001 — ENA-001 will be prepared in Ringer's lactate solution. A loading dose will be administered for 20 minutes followed by continuous infusion until the patient meets the criteria for PACU discharge (≥ 9 Aldrete score) or ABG reveals PaCO2 < 30 mmHg with pH in the normal range. ENA-001 is for IV injection ready for use per subject by the investigational pharmacy, according to the randomization schedule.

SUMMARY:
This study is a Phase II, randomized, placebo-controlled, double-blind trial in 200 subjects having general anesthesia for major elective surgery with postoperative pain management to evaluate the efficacy, safety and tolerability of ENA-001 as a therapy to prevent post operative respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give written informed consent for the trial and willing/able to adhere to study procedures.
2. Scheduled to undergo a major elective surgery, including abdominal, laparoscopic, nephrology, thoracic (non-cardiac), orthopedic (e.g., shoulder and ankle surgery), where the subject will be transferred to recover in the general postanesthesia recover unit (PACU) and extubation will be performed in the operating room or PACU.
3. Undergoing surgical procedure with a intraoperative requirement of ≥ 250 µg of fentanyl; Enrolled base on expected pain management to necessitate ≥ 250 µg of fentanyl intraoperatively.
4. Male and female, ≥18 years of age.
5. American Society of Anesthesiologists (ASA) physical status classification 1-3.
6. Have no clinical or electrocardiographic signs of ischemic heart disease as determined by the Investigator. The Screening 12 lead ECG conduction intervals must be within gender specific normal range (e.g., QTcF female &lt; 450 msec QTcF males &lt; 430 msec, PR interval ≤ 220 msec). ECGs are to be judged by the investigator or sub-investigator as per standardized procedures.
7. Clinical laboratory tests (blood hematology, blood chemistry, coagulation and urinalysis) must not include any significant clinical abnormalities.
8. Vital sign measurements must be within the following ranges during screening and on the day of dosing:

   1. body temperature, ≥35.5°C to ≤37.5°C
   2. systolic blood pressure, ≥90 to ≤150 mm Hg
   3. diastolic blood pressure, ≥50 to ≤95 mm Hg
   4. pulse rate, ≥40 to ≤100 bpm
9. Non-vasectomized men must agree to use a condom with spermicide, double-barrier contraception, abstain from heterosexual intercourse, or have a sole-sexual partner of non childbearing potential during the trial and for 3 months after stopping the medication. Male subjects must agree not to donate sperm from the time of dosing until 90 days after dosing.
10. Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative pregnancy test prior to enrolment and must agree to the following contraception requirements from screening through 3 months after dosing of the study drug:

    1. Be sexually inactive (abstinent)
    2. Intrauterine device in place for at least three months prior to dosing with a barrier method (condom or diaphragm) and spermicide throughout the study.
    3. Double barrier methods (e.g., condom and diaphragm) with spermicide for at least 14 days prior to dosing and throughout the study.
    4. Surgical sterilization of the partner (vasectomy at least six months prior to dosing) with a barrier method (e.g., condom or diaphragm) and spermicide throughout the study.
    5. Female subjects who claim to be sexually inactive but become sexually active during the course of the study must agree to use a double barrier method (e.g., condom and diaphragm) with spermicide from the time of the start of sexual activity through completion of the study. In addition, female subjects of childbearing potential must be advised to remain sexually inactive or to keep the same birth control method for at least 14 days following study medication administration. Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to dosing:

    <!-- -->

    1. Hysteroscopic sterilization and be using a barrier method (e.g., condom or diaphragm) and spermicide throughout the study.
    2. Bilateral tubal ligation or bilateral salpingectomy and be using a barrier method (e.g., condom or diaphragm) and spermicide throughout the study.
    3. Hysterectomy.
    4. Bilateral oophorectomy. Women with amenorrhea for at least 1 year prior to dosing and who have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status, are considered post menopausal and therefore of non-childbearing potential.
11. Subjects must be free of any clinically significant disease that would interfere with the study evaluations.

Exclusion Criteria:

1. Ongoing treatment for a pre-existing chronic pain condition
2. Use of an epidural / spinal block / major nerve block for the surgical procedure
3. Surgical procedure that may interfere with the collection of data under the study protocol, such as craniofacial surgery which may impact the placement of a face mask for pulmonary function measurements.
4. Current diagnosis of psychiatric disease, including anxiety disorder, that is uncontrolled and/or restricting normal daily function.
5. History of alcohol abuse (more than an average of 2-drinks per day) within the past 2 years.
6. History of drug abuse within the past 2 years.
7. History of regular smoking within the past year (>5 per week means exclusion).
8. Positive for HIV, or Hepatitis B or C at screening.
9. Blood donation or blood loss within 60 days of screening or plasma donation within 7 days of screening.
10. Current or recent presentation of clinically significant of dyspnea, asthma, tuberculosis, chronic obstructive pulmonary disease, sleep apnea (central or obstructive) or any other ventilatory / lung disease.
11. Treatment with another investigational drug within 3 months prior to screening or having participated in more than four investigational drug studies within 1 year prior to screening.
12. History of moderate to severe motion sickness.
13. Subjects who are unwilling to remove excessive facial hair preventing sealing of the occlusive face mask.
14. Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
15. Any surgical or medical condition which might significantly alter the distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following, and be discussed with the sponsor prior to enrollment into the trial:

    1. history of pancreatic injury or pancreatitis;
    2. history or presence of liver disease or liver injury;
    3. history or presence of impaired renal function as indicated by clinically significant elevation in creatinine, BUN/urea, urinary albumin, or clinically significant urinary cellular constituents; or
    4. history of urinary obstruction or difficulty in voiding.
16. Subject who has a history of any infectious disease within 4 weeks prior to drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial.
17. Subjects who are part of the study staff personnel or family members of the study staff personnel.
18. Subjects who have demonstrated allergic reactions (e.g., food, drug, atopic reactions or asthmatic episodes) which, in the opinion of the investigator and sponsor, interfere with their ability to participate in the trial.
19. Subjects who have a history of malignancy and are in remission <5 years.
20. Personal or family history of malignant hyperthermia.
21. History of arrhythmias or ECG conductance abnormalities.
22. Subjects with history of known difficult airway access and presence of a "non-reassuring" airway exam (as determined by the investigator), gastroesophageal reflex disease, gastric motility disorders, or delayed gastric emptying, or any condition that may lead to delayed gastric emptying such as diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of ENA-001 on pulmonary ventilation when administered to 100 subjects via continuous infusion of a loading dose of 2.0 mg/kg/hr for 20 minutes followed by a maintenance dose of 1.1 mg/kg/hr | 2 hours
  To evaluate the effect of ENA-001 on pulmonary ventilation following extubation/airway removal up to two hours beyond cessation of treatment. Endpoint is arterial CO2 tension (PaCO2)

IPD SHARING:
Plan to Share IPD: No